CLINICAL TRIAL: NCT06752785
Title: Clinical Study on the Safety and Efficacy of CD19/CD22 CAR-T Cell Therapy in MRD-Positive B-lineage Acute Lymphoblastic Leukemia in Children.
Brief Title: CD19/CD22 CAR-T Cell Therapy in MRD-Positive B-lineage Acute Lymphoblastic Leukemia in Children.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024423A01
Record Dates: First submitted 2024-12-12; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: B-ALL, CAR-T
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRD-Positive B-lineage Acute Lymphoblastic Leukemia (Experimental): Children of MRD-Positive B-lineage Acute Lymphoblastic Leukemia; CD19/CD22 CAR-T
  Interventions: Drug: CAR-T Therapy

INTERVENTIONS:
Drug: CAR-T Therapy — CD19/CD22 CAR-T cell therapy

SUMMARY:
In this study, CD19/CD22 dual-target CAR-T therapy will be carried out among children patients who are still positive after induction remission, and subsequent chemotherapy will continue after CAR-T cells exert their functions. This study intends to use retroviral vector-based tandem CAR-T cells targeting CD19/CD22 to treat MRD-positive ALL. The CAR-T cells were provided by Shenzhen Cell Valley. The results of the research team from Stanford University School of Medicine in the United States have already demonstrated the feasibility and safety of producing bispecific CD19/CD22.BB.z-CAR T cells in a closed system as well as the high clinical activity shown in the treatment of CAR19-resistant B-ALL (B-lineage acute lymphoblastic leukemia) and LBCL (Large B-cell lymphoma). The investigators look forward to expanding the application of CAR-T cells in MRD positive B-ALL through this clinical study on safety and efficacy and greatly improving the prognosis of children patients with this type of B-ALL.

DETAILED DESCRIPTION:
This clinical trial is a single-center, open-label, single-arm clinical trial to evaluate the safety and efficacy of CAR-T cell treatment for MRD-positive B-ALL. The specific trial process is divided as follows:

1. Screen the enrolled population to determine the indications and exclusion criteria for cell treatment. In brief, intermediate-risk patients with positive MRD on day 46 of induction through flow cytometry according to CCCG-ALL regimen.
2. Sign the informed consent form.
3. CAR-T cell preparation: collect autologous lymphocytes and produce CAR-T cells targeting the CD19/CD22 target.
4. Lymphocyte depletion pretreatment: according to the patient's condition, select the FC regimen (fludarabine 30 mg/m²/day for 4 days; cyclophosphamide 500 mg/m²/day for 2 days) before autologous transplantation.
5. Cell intravenous infusion: dose: 3 × 10⁶/kg (allowable fluctuation range: 2 × 10⁶/kg - 4 × 10⁶/kg). Obeserve adverse reactions including CRS and ICANS.
6. Evaluate the efficacy after the first cell infusion by MRD test .
7. Continue chemotherapy after one month of CART according CCCG-ALL regimen from the second high-dose MTX of consolidation stage.
8. Follow-up after the completion of the clinical study: within the first month after cell infusion, the subject needs to complete the relevant examinations required for follow-up on the 7th, 14th, 21st, and 30th days. Depending on the patient's condition, the number of detections may also be increased; from the 2nd to 6th months after infusion, follow-up once a month; from 6 months to 2 years after infusion, follow-up once every 3 months. From 2 to 5 years after infusion, follow-up once a year. After that, enter long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Parents or legal guardians fully understand, are informed of this study and sign the informed consent form (ICF); are willing to follow and can complete all test procedures.
2. Chinese children aged 1-18 years old at the time of screening, regardless of gender, with a body weight ≥ 10 kg.
3. Bone marrow examination confirms that MRD is still positive on the 46th day after induction remission.
4. Tumor cells in the bone marrow (BM) or peripheral blood (PB) express CD19/CD22 within 3 months before screening.
5. Good organ function, which needs to meet the following criteria: (1)ALT ≤ 5 times the upper limit of normal value (ULN); (2)total bilirubin ≤ 2 times ULN (Gilbert's syndrome ≤ 3 times ULN); (3)without > grade 1 dyspnea when not inhaling oxygen, and oxygen saturation > 95%; (4)left ventricular ejection fraction (LVEF) ≥ 50%; (5)serum creatinine ≤ 1.5 times ULN.
6. Karnofsky score (≥ 16 years old) ≥ 70 or Lansky (< 16 years old) score ≥ 50.
7. Expected survival period of at least 12 weeks.
8. Have sufficient venous access (for apheresis or venous blood sampling), and have no other contraindications for blood cell separation.

Exclusion Criteria:

1. Have genetic diseases, except Down syndrome.
2. Have a history of other malignancies or have other malignancies simultaneously.
3. Meet any of the following conditions: (1)hepatitis B surface antigen (HBsAg) positive or HBV DNA quantification higher than the upper limit of normal value; (2)hepatitis C antibody (HCV Ab) positive and HCV RNA quantification higher than the upper limit of normal value; (3)human immunodeficiency virus antibody (HIV-Ab) positive; (4)Treponema pallidum antibody (TP-Ab) positive; (5)EBV DNA higher than the upper limit of normal value; (6)cytomegalovirus DNA higher than the upper limit of normal value.
4. Have or are suspected to have uncontrolled or require intravenous drug treatment for fungal, bacterial, viral or other infections.
5. Long-acting G-CSF is prohibited within 21 days before screening, and short-acting G-CSF is prohibited within 7 days before screening.
6. Have active central nervous system leukemia.
7. Are allergic to albumin and aminoglycoside antibiotics.
8. Have undergone organ transplantation (except hematopoietic stem cell transplantation).
9. Have participated in other interventional clinical studies within 3 months before screening (received active test drug treatment), or intend to participate in another clinical trial or receive anti-tumor treatment other than that specified in the protocol during the entire study period.
10. Cannot tolerate chemotherapy and cytokine storm due to impaired function of important organs.
11. Other situations that the investigator deems not suitable for participating in this clinical trial.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Validity exploration | One year after CAR-T treatment
  According to the efficacy evaluation criteria for ALL in the "NCCN Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (2024.V5)", the complete remission(CR) rate will be evaluated at 1 year after CAR-T treatment.CR is generally measured in percentage(%).

CONTACTS AND LOCATIONS:
Overall Officials: Hua Jiang, phd, Study Director — Guangzhou Medical University Affiliated Women and Children's Medical Center
Locations (1):
- Guangzhou Medical University Affiliated Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Researchers or funders may have conflicts of interest.

REFERENCES:
- [Background] Cordoba S, Onuoha S, Thomas S, Pignataro DS, Hough R, Ghorashian S, Vora A, Bonney D, Veys P, Rao K, Lucchini G, Chiesa R, Chu J, Clark L, Fung MM, Smith K, Peticone C, Al-Hajj M, Baldan V, Ferrari M, Srivastava S, Jha R, Arce Vargas F, Duffy K, Day W, Virgo P, Wheeler L, Hancock J, Farzaneh F, Domning S, Zhang Y, Khokhar NZ, Peddareddigari VGR, Wynn R, Pule M, Amrolia PJ. CAR T cells with dual targeting of CD19 and CD22 in pediatric and young adult patients with relapsed or refractory B cell acute lymphoblastic leukemia: a phase 1 trial. Nat Med. 2021 Oct;27(10):1797-1805. doi: 10.1038/s41591-021-01497-1. Epub 2021 Oct 12. PMID 34642489
- [Background] Wang T, Tang Y, Cai J, Wan X, Hu S, Lu X, Xie Z, Qiao X, Jiang H, Shao J, Yang F, Ren H, Cao Q, Qian J, Zhang J, An K, Wang J, Luo C, Liang H, Miao Y, Ma Y, Wang X, Ding L, Song L, He H, Shi W, Xiao P, Yang X, Yang J, Li W, Zhu Y, Wang N, Gu L, Chen Q, Tang J, Yang JJ, Cheng C, Leung W, Chen J, Lu J, Li B, Pui CH. Coadministration of CD19- and CD22-Directed Chimeric Antigen Receptor T-Cell Therapy in Childhood B-Cell Acute Lymphoblastic Leukemia: A Single-Arm, Multicenter, Phase II Trial. J Clin Oncol. 2023 Mar 20;41(9):1670-1683. doi: 10.1200/JCO.22.01214. Epub 2022 Nov 8. PMID 36346962
- [Background] Pan J, Tang K, Luo Y, Seery S, Tan Y, Deng B, Liu F, Xu X, Ling Z, Song W, Xu J, Duan J, Wang Z, Li C, Wang K, Zhang Y, Yu X, Zheng Q, Zhao L, Zhang J, Chang AH, Feng X. Sequential CD19 and CD22 chimeric antigen receptor T-cell therapy for childhood refractory or relapsed B-cell acute lymphocytic leukaemia: a single-arm, phase 2 study. Lancet Oncol. 2023 Nov;24(11):1229-1241. doi: 10.1016/S1470-2045(23)00436-9. Epub 2023 Oct 17. PMID 37863088
- [Background] Buechner J, Caruana I, Kunkele A, Rives S, Vettenranta K, Bader P, Peters C, Baruchel A, Calkoen FG. Chimeric Antigen Receptor T-Cell Therapy in Paediatric B-Cell Precursor Acute Lymphoblastic Leukaemia: Curative Treatment Option or Bridge to Transplant? Front Pediatr. 2022 Jan 25;9:784024. doi: 10.3389/fped.2021.784024. eCollection 2021. PMID 35145941
- [Background] Pui CH, Yang JJ, Hunger SP, Pieters R, Schrappe M, Biondi A, Vora A, Baruchel A, Silverman LB, Schmiegelow K, Escherich G, Horibe K, Benoit YC, Izraeli S, Yeoh AE, Liang DC, Downing JR, Evans WE, Relling MV, Mullighan CG. Childhood Acute Lymphoblastic Leukemia: Progress Through Collaboration. J Clin Oncol. 2015 Sep 20;33(27):2938-48. doi: 10.1200/JCO.2014.59.1636. Epub 2015 Aug 24. PMID 26304874
- [Background] Pui CH, Yang JJ, Bhakta N, Rodriguez-Galindo C. Global efforts toward the cure of childhood acute lymphoblastic leukaemia. Lancet Child Adolesc Health. 2018 Jun;2(6):440-454. doi: 10.1016/S2352-4642(18)30066-X. Epub 2018 Mar 30. PMID 30169285